CLINICAL TRIAL: NCT01133080
Title: Minocycline as an Adjunctive Therapy for Schizophrenia: a Randomized Controlled Study
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shalvata Mental Health Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SHA-0008-10
Record Dates: First submitted 2010-05-26; First posted 2010-05-28 (Estimated); Last update posted 2012-01-05 (Estimated); Status verified 2012-01

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Minocycline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Minocycline (Experimental)
  Interventions: Drug: Minocycline
- Placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Minocycline — minocycline 200 mg/day orally in two divided doses for the second week. From weeks 3 to weeks 5, minocycline 400 mg/day orally in two divided doses.
  Arms: Minocycline
Drug: placebo — placebo 200 mg/day orally in two divided doses for the first week. placebo 200 mg/day orally in two divided doses for the second week.
  From weeks 3 to weeks 5, placebo 400 mg/day orally in two divided doses.
  Arms: Placebo

SUMMARY:
Double - Blind, Randomized, single centered study. The purpose of this study is to assess the feasibility of minocycline vs. placebo, added to atypical antipsychotic medications, for positive symptoms in adults suffering from schizophrenia.

ELIGIBILITY:
Inclusion Criteria:

* Men and women 20-65 years of age.
* Primary DSM-IV diagnosis of Schizophrenia based on SCID for schizophrenia and confirmed by two senior psychiatrists.
* Patients who scored "moderate" (4) or higher on at least three of seven positive items in PANSS
* Initiated on treatment with atypical anti-psychotic medication.
* Capable and willing to provide informed consent
* Able to adhere to the treatment schedule
* Able to read, hear, write and speak the local language.
* Has signed a written informed consent to participate in the study

Exclusion Criteria:

* Patients with acute, unstable, significant, or untreated medical illness besides schizophrenia including alcohol and drug dependence, or depression.
* Current suicidal ideation or history of a suicide attempt in the past 3 years
* Known or suspected pregnancy or women of childbearing potential and not using a medically accepted form of contraception when engaging in sexual intercourse. or women who are breastfeeding
* Subjects who were taking a known contraindication to minocycline treatment.
* Subjects who had received treatment with minocycline or β-lactam antibiotics in the preceding half year before study entry.
* Subjects who were under compulsory hospitalization.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2010-06; Primary Completion 2013-01 (Estimated); Study Completion 2013-01 (Estimated)

PRIMARY OUTCOMES:
Positive symptoms | from baseline to the end of the study (day 56)
  Positive symptoms: The change in Scale for the Positive and Negative Syndrome Scale (PANSS) score from baseline to the end of the study and the change in Clinical Global Impression Scale (CGI).

CONTACTS AND LOCATIONS:
Overall Officials: Yechiel Levkovitz, MD, PhD, Principal Investigator — Shalvata MHC
Locations (2):
- Israel (2):
  - Shalvata Mental Health Center, Hod HaSharon
  - shalvata MHC, Hod HaSharon